CLINICAL TRIAL: NCT03048565
Title: An Exploratory Randomised Pilot Trial Examining the Potential Effectiveness of an Online Mindfulness Based Stress Reduction Programme for Informal Caregivers of People With Chronic Illnesses.
Brief Title: A Trial of an Online Mindfulness Based Programme for Informal Caregivers of People With Chronic Illnesses
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment challenges
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: Family Carers Ireland (Unknown)
Responsible Party: Principal Investigator, Margarita Corry, Assistant Professor, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12
Record Dates: First submitted 2017-02-06; First posted 2017-02-09 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Chronic Illness
Keywords: mindfulness; caregivers
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): No intervention
- Mindfulness based Stress Reduction (Experimental): This is an active intervention The MBSR programme is delivered online with weekly telephone and email contact from a trained mindfulness teacher. Participants are encouraged to practice mindfulness exercises and homework between sessions. The online programme was developed be a trained mindfulness teacher.
  Interventions: Behavioral: MBSR

INTERVENTIONS:
Behavioral: MBSR — Mindfulness is a skill that helps people manage their thoughts so that the stressful impact of unhelpful thoughts can be limited. The aim of the mindfulness based intervention in this study is to help caregivers manage stressful thoughts and events and help them respond to life stressors in a positive way.
  Arms: Mindfulness based Stress Reduction

SUMMARY:
This is a pilot feasibility study testing a mindfulness based intervention with caregivers of people with chronic illnesses

DETAILED DESCRIPTION:
The primary aim of the project is to pilot test the delivery of an online Mindfulness Based Stress Reduction (MBSR) programme to informal caregivers of people with chronic illnesses in one region in Ireland so as to determine the feasibility of delivering the intervention to caregivers in Ireland.

A two-group randomised pilot-feasibility trial comparing the online MBSR programme (intervention) with no programme (control). The MBSR programme is delivered online over 8 weeks. Weekly email and telephone contact will be maintained with participants in the intervention group for the duration of the delivery of the intervention. Participants are encouraged to practice mindfulness exercises and homework between sessions. The online programme was developed by a trained mindfulness teacher and a mindfulness teacher will conduct the weekly email and telephone call to participants in the intervention group. The study sample are caregivers in the Dublin region who are members of Family Carers' Ireland. A total of 80 caregivers will be recruited to the study, 40 per group, based on 1:1 randomisation using a computer-randomised number generator.

Baseline (pre-intervention) and post intervention participant outcome data (stress, mindfulness and QoL) will be collected using self-reported validated scales administered to participants by post, with stamped-addressed envelopes provided for return. Other pilot measures (i.e. study processes) will be monitored and assessed by the research team to determine potential refinement needs. Feasibility outcome data will be collected by the research team (including time to recruit, attendance at classes, willingness of participants to be randomised) and by the participants (expenses diary) during the study period, using predesigned data collection forms. Mean differences with 95% confidence intervals will be calculated to determine any significant differences between the groups on the outcomes of stress, mindfulness and QoL.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age and over
* Provide unpaid care to an adult or child with a chronic illness
* Not suffer from a severe mental illness
* Be ready to commit to the course at this point in their lives.

Exclusion Criteria:

* Caregivers who are under the age of 18 years.
* Caregivers who have a serious mental illness, such as severe anxiety/depression.
* Caregivers who are in receipt of current and regular treatment from a psychologist or psychiatrist.
* Caregivers with an active or recent physical addiction to alcohol or drugs.
* Caregivers who are already engaged in similar research.
* Caregivers who have already participated in mindfulness based stress reduction (MBSR) or MBCT training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2017-10-04 (Actual); Study Completion 2017-10-04 (Actual)

PRIMARY OUTCOMES:
Change over time in Calgary Symptoms of Stress Inventory (C-SOSI) | up to 2 weeks and 6 months post-intervention
  Response to stressful situations
Change over time in Perceived Stress Scale | up to 2 weeks and 6 months post-intervention
  perceived stress
Change over time in Cognitive and Affective Mindfulness Scale Revised (CAMS-R) | up to 2 weeks and 6 months post-intervention
  Mindfulness
Change over time in The Adult Carer Quality of Life Questionnaire | up to 2 weeks and 6 months post-intervention
  Quality of Life

OTHER OUTCOMES:
Caregiver MBCT Programme Evaluation Form | up to 2 weeks post-intervention
  programme evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Corry, Principal Investigator — University of Dublin, Trinity College
Locations (2):
- Ireland (2):
  - Trinity College Dublin, Dublin
  - Trinity College Dubliln, Dublin

IPD SHARING:
Plan to Share IPD: Undecided